CLINICAL TRIAL: NCT04880044
Title: Detection of Barrett s Esophagus in Patients Without Gastroesophageal Reflux Disease (GERD) Symptoms
Brief Title: Detection of Barrett s Esophagus in Patients Without GERD Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CASE1221
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EC/EG & EGD (Experimental): Participants will complete a study questionnaire about reflux symptoms. Performance of an EsoCheck (EC) procedure; the EC sample will subsequently be tested with the EsoGuard (EG) assay
  If EG assay results come back positive, participant is requested to complete standard of care (SOC) upper endoscopy (tissue samples collected)
  If EG assay results come back negative, selected participants (100 volunteers) will also undergo a research EGD if they consent
  Interventions: Diagnostic Test: EsoCheck/EsoGuard (EC/EG); Diagnostic Test: Esophago-gastro-duodenoscopy (EGD)

INTERVENTIONS:
Diagnostic Test: EsoCheck/EsoGuard (EC/EG) — EC is a swallowed capsule on a tethered catheter that obtains a touch sample of the distal esophagus. The obtained sample is placed in a buffer and sent to a diagnostics lab for testing of methylated markers from extracted DNA. EG is a methylated DNA test . A positive EG is associated with Barrett's esophagus at all its stages.
Diagnostic Test: Esophago-gastro-duodenoscopy (EGD) — SOC diagnostic endoscopic procedure that visualizes the upper part of the gastrointestinal tract down to the duodenum. Tissue samples collected.

SUMMARY:
The purpose of this study is to develop a method to detect Barrett's esophagus (BE) in individuals with a new office-based diagnostic test.

DETAILED DESCRIPTION:
This study will investigate whether using EsoCheck/EsoGuard(EC/EG) can detect BE in individuals at risk for BE who are currently not being detected and are not undergoing routine esophago-gastro-duodenoscopy (EGD)

BE can only be diagnosed by performing upper endoscopy. Up to 500 adults who have risk factors for BE but do not have chronic heartburn or regurgitation will be enrolled in this study. This will include the EsoCheck/EsoGuard determination along with the upper endoscopy for qualifying EsoGuard negative subjects

ELIGIBILITY:
Inclusion Criteria:

* No known coagulopathy, no known esophageal varices.
* No significant dysphagia or odynophagia
* Absence of chronic GERD, defined as five or more years of heartburn or regurgitation with symptoms at least once a week when not on medications for GERD symptoms.
* Subjects to qualify must meet criterion 3, be over age 50, and have two additional risk factors for BE (white race, central obesity defined as waist size >35 inches for women and >40 inches for men, male gender, current smoker or smoking history >10 pack years, confirmed family history in at least two members with one being a first degree relative).

Exclusion Criteria:

* History of prior EGD procedure
* Inability to provide written informed consent
* History of weekly of more frequent heartburn or regurgitation for five or more years
* On anti-coagulant drug(s)that cannot be temporarily discontinued or coagulopathy with international normalized ratio (INR) > 1.5
* Known history of esophageal varices or esophageal stricture
* Any contraindication, as deemed inInvestigator's medical judgment, to undergoing the EsoCheck procedure, undergoing the EGDprocedure,and/or having biopsies taken, including but not limited to due to comorbidities such as coagulopathy or a known history of esophageal diverticula, esophageal fistula and/or esophageal ulceration
* History of difficulty swallowing (dysphagia) or painful swallowing (odynophagia), including swallowing pills
* Oropharyngeal tumor
* History of esophageal or gastric surgery, with exception on uncomplicated surgical fundoplication procedure
* History of myocardial infarction or cerebrovascular accident within past 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Positive predictive value (PPV) of EC/EG in a non-GERD population that has three or more non-GERD risk factors for BE. | Up to 2 months
  PPV of EC/EG in a non-GERD population that has three or more non-GERD risk factors for BE. Participants who are at risk will be offered EC/EG. Those who are positive will undergo subsequent EGD
  PPV = (EC/EG positive & EGD positive) / ((EC/EG positive & EGD positive) + (EC/EG positive & EGD negative))
Proportion of participants negative via EC/EG who subsequently are proven negative via EGD | Up to 2 months
  Negative Predictive Value (NPV):
  Proportion of participants negative via EC/EG who subsequently are proven negative via EGD. This will be measured by offering EGD to a proportion of patients who are EC/EG negative.

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Chak, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that result in publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Derived] Chak A, Keerthy K, Wang GM, Brock W, Bednarchik B, Guptha R, Verma S, Moinova H, Tatsuoka C, Dumot J, Thomas S, Willis JE, Markowitz S. Nonendoscopic Detection of Barrett's Esophagus on Patients Without Gastroesophageal Reflux Disease Symptoms. Am J Gastroenterol. 2026 Jan 1;121(1):258-261. doi: 10.14309/ajg.0000000000003669. Epub 2025 Aug 1. PMID 40748349